CLINICAL TRIAL: NCT01473628
Title: Randomized Trial of Radiation Therapy With and Without Rituximab for Patients With Stage I II Follicular Lymphoma Grade I/II
Brief Title: Radiation Therapy and Rituximab in Treating Patients With Stage I-II Grade 1 or Grade 2 Follicular Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0283; NCI-2012-00734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0283 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Ann Arbor Stage I Grade 1 Follicular Lymphoma; Ann Arbor Stage I Grade 2 Follicular Lymphoma; Ann Arbor Stage II Grade 1 Follicular Lymphoma; Ann Arbor Stage II Grade 2 Follicular Lymphoma
MeSH Terms: interventions — Watchful Waiting; Observation; Radiotherapy; Radiation; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (radiation therapy and rituximab) (Experimental): Patients undergo radiation therapy five days a week for 2.5 weeks (12 treatments) and receive rituximab IV over 4-6 hours weekly with the start of radiation for 4 weeks and then every 2 months for up to 4 additional doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation Therapy; Biological: Rituximab
- Arm II (radiation therapy and observation) (Experimental): Patients undergo radiation therapy five days a week for 2.5 weeks and then undergo observation.
  Interventions: Other: Clinical Observation; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Clinical Observation — Undergo observation
  Other Names: observation
  Arms: Arm II (radiation therapy and observation)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
  Arms: Arm I (radiation therapy and rituximab)

SUMMARY:
This randomized phase I/II trial studies radiation therapy and rituximab in treating patients with stage I-II grade 1 or grade 2 follicular lymphoma. Radiation therapy uses high energy x-rays to kill cancer cells. Immunotherapy with monoclonal antibodies, such as rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving radiation therapy with rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if rituximab concurrently with radiation followed by maintenance rituximab offers a superior benefit over radiation alone. Specifically looking at the progression free survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo radiation therapy five days a week for 2.5 weeks (12 treatments) and receive rituximab intravenously (IV) over 4-6 hours weekly with the start of radiation for 4 weeks and then every 2 months for up to 4 additional doses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo radiation therapy five days a week for 2.5 weeks and then undergo observation.

After completion of study treatment, patients are followed up at 3 and 6 months, every 6 months for 2 years, yearly for 3 years, and then every 2 years for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with stage I and II follicular lymphoma, pathologically confirmed at MD Anderson Cancer Center (MDACC) to be grade 1 or 2
* Prophylactic use of lamivudine in patients that have antibody positive (+), but no active infection will be up to the treating physician
* Absolute neutrophil count (ANC) >= 1000/mm^3; this value must be obtained within four weeks before protocol entry
* Platelets >= 80,000/mm^3; this value must be obtained within four weeks before protocol entry
* Hemoglobin >= 8 g/dL; this value must be obtained within four weeks before protocol entry
* Bilirubin =< 1.5 times the upper limit of normal (ULN); this value must be obtained within four weeks before protocol entry
* Alanine aminotransferase (ALT) =< 2 times the ULN or aspartate aminotransferase (AST) =< 2 times the ULN; these values must be obtained within four weeks before protocol entry
* Performance status >= 2
* Patients are required to have adequate renal function as indicated by a serum creatinine =< 2.5 mg/dL; this value must be obtained within four weeks before protocol entry
* No prior known allergic reaction to monoclonal antibodies
* Male patients must agree to use a barrier method of contraception or agree to abstain from heterosexual activity for the duration of the study
* Female patients must be willing to use two adequate barrier methods of contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study or be post menopausal (free from menses > two years or surgically sterilized)
* Female patients of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [B HCG]) within 72 hours of receiving the first dose of rituximab
* Patients must have the ability able to give informed consent

Exclusion Criteria:

* Patients with active hepatitis B and/or hepatitis C infection
* Patients with known human immunodeficiency virus (HIV) infection
* Patients with active infections requiring specific anti-infective therapy are not eligible until all signs of infections are resolved
* Patients who had previous radiation dose to the site of the current primary disease, which would lead to violation of known radiation tolerance limit of that particular site if treated again
* Patients with pre-existing cardiovascular disease requiring ongoing treatment; this includes: congestive heart failure III/IV as defined by New York Heart Association (NYHA); uncontrolled cardiac arrhythmia; unstable angina pectoris; and recent myocardial infarction (MI) (within 6 months)
* Patients who are pregnant or breast-feeding
* Patient with concurrent use of complementary or alternative medicines
* Patients with psychiatric illness and/or social situations that would limit compliance with the study medication and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-05-20 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that remain progression free, defined as progressive disease or death due to disease | Up to 15 years
  The student t-test or the Wilcoxon rank sum test will be used to compare continuous variables between two different patient groups. The chi-square test or the Fisher's exact test will then be applied to assess the association between two categorical variables. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate. Kaplan-Meier survival curves will also be constructed.

SECONDARY OUTCOMES:
Overall survival | Up to 15 years
  Estimated using the Kaplan-Meier method. The log-rank test will be performed to test the difference in time-to-event distributions between patient groups. The Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis.
Progression free survival rate | Up to 15 years
  Estimated using the Kaplan-Meier method. The log-rank test will be performed to test the difference in time-to-event distributions between patient groups. The Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina S Dabaja, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org